CLINICAL TRIAL: NCT05952362
Title: The Effect of Smartphone Addiction and Mental Fatigue on Working Memory in University Students
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/07-08
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-07

CONDITIONS: Smartphone Addiction; Mental Fatigue
Keywords: working memory; mental fatigue; smartphone addiction
MeSH Terms: conditions — Internet Addiction Disorder; Mental Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the effects of smartphone addiction and mental fatigue on working memory in university students.

DETAILED DESCRIPTION:
University students who meet the inclusion and exclusion criteria will be informed about the study and the participants who agree to participate in the study will be given the Turkish version of "Smartphone Addiction Scale", ''Mental Fatigue Scale'' and "Working Memory Questionnaire" tests, respectively. 120 university students will included in the study. To evaluate between correlation of tests will used to correlation analysis tests. In addition, it will be investigated whether there is a difference between 1.2.3 and 4th grades in terms of Smartphone Addiction, Mental Fatigue Scale and Working Memory Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Being a university student
* Be between the ages of 18-25
* Using a smartphone for at least one hour a day

Exclusion Criteria:

* Having musculoskeletal pain
* Having had surgery in the last 6 months
* Decline to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 120 university students
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Working Memory Questionnaire | Baseline (First assessment)
  The Working Memory Questionnaire (WMQ) is a self-administered scale proposed by Vallat-Azouvi. It assesses the three different working memory domains (memory storage, attention, and executive functions). It consists of 30 questions, each scored on a five-point Likert-type scale ranging from 0 (not at all) to 4 (extremely). The total score varies between 0 and 120. Higher scores represent more memory difficulties/complaints.

SECONDARY OUTCOMES:
Smartphone Addicition Scale-Short Version | Baseline (First assessment)
  This instrument to examine smartphone addiction was developed by Kwon et al. This scale consisted of six factors with ten items each, rated using the six-point Likert scale (1: strongly disagree, 2: disagree, 3: weakly disagree, 4: weakly agree, 5: agree, and 6: strongly agree).
Mental Fatigue Scale | Baseline (First assessment)
  The Mental Fatigue Scale (MFS) is a 15-item questionnaire that specifically evaluates mental fatigue. It includes affective, cognitive and sensory symptoms, duration of sleep and daytime variation in symptom severity. It has a 7-point Likert-type scale and is scored between 0 and 3. A rating of 0 indicates normal function, 1 slight problem, 2 significant problems and 3 maximum problems. There are also items such as 0.5, 1.5, 2.5 for marking when individuals fall between 2 items (0.5, 1.5, 2.5). The total score of the scale is obtained by summing the scores of the first 14 questions. The last question is evaluated as yes or no. The scores range from 0 to 42 and 0-10 indicates no mental fatigue problem, 10.5-14.5 indicates slight mental fatigue, 15-20 indicates fairly serious mental fatigue, and ≥ 20.5 indicates serious mental fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye AKKURT, PhD, Study Director — Kutahya Health Sciences University; Cihan Caner AKSOY, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)